CLINICAL TRIAL: NCT03042520
Title: Long-term Hepatic and Extra-hepatic Outcomes of Chronic Hepatitis C Patients Post Sofosbuvir-based Interferon-free Treatment (LONGHEAD Study)
Brief Title: Long-term Outcomes of Chronic Hepatitis C Patients Post Sofosbuvir-based Treatment
Acronym: LONGHEAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other); National Taiwan University Hospital (Other); National Cheng-Kung University Hospital (Other); Chi Mei Medical Hospital (Other); China Medical University, China (Other); Mackay Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Changhua Christian Hospital (Other); Pusan National University Hospital (Other); Asan Medical Center (Other); Korea University (Other); Inje University (Other); Korea University Guro Hospital (Other); Kyungpook National University Hospital (Other); Seoul National University Hospital (Other); Severance Hospital (Other); Samsung Medical Center (Other); Seoul National University Bundang Hospital (Other); Soon Chun Hyang University (Other); Seoul St. Mary's Hospital (Other); Gachon University Gil Medical Center (Other); Dong-A University Hospital (Other); Gangnam Severance Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: irb20160082
Record Dates: First submitted 2016-12-21; First posted 2017-02-03 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Liver Fibroses; HepatoCellular Carcinoma; Cryoglobulinemia; Metabolic Disease; Diabetes Mellitus
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Cryoglobulinemia; Metabolic Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IFN-based therapy historical controls: Patients who had ever participated the parent studies, GS-US-334-0115 or GS-US-337-0131, will be invited to participate the current study in outpatient clinic. For the patients who have participated study will be invited to participate the current study as matched historical control n our outpatient clinic,
  Interventions: Other: Observation only
- Sofosbuvir-based therapy observational group: 1. Patients ≥ 20 of years who had ever participated in parent studies, GS-US-337-0131 (NCT02021656) or GS-US-334-0115 (NCT02021643)
  2. Patients who had received at least one dose of sofosbuvir-based therapy in the parent studies.
  Who IFN-based therapy historical controls, matched with sex, age, level of liver fibrosis and virological response:
  1. Patients ≥ 20 of years who had received peginterferon plus ribavirin therapy with match of sex, age, level of liver fibrosis and virological response
  2. Patients who have ever participated study will be collected as historical control.
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only

SUMMARY:
Primary Objective:

To evaluate the long-term outcomes including liver related morbidity, mortality and hepatocellular carcinoma (HCC) development as compared to those of historical control with interferon(IFN)-based treatment.

Secondary Objective:

1. To access liver fibrosis progression/regression in CHC patients after sofosbuvir-based treatment.
2. To investigate the long-term outcomes of extrahepatic manifestations of the sofosbuvir-based treated cohort as compared to their pretreatment status.

DETAILED DESCRIPTION:
Primary Endpoint:

To evaluate the long-term event-free effect after sofosbuvir-based therapy, in terms of free of major liver events (including HCC, decompensation with ascites, variceal bleeding, hepatic encephalopathy, and liver-related mortality) in CHC patients.

Secondary Endpoints:

1. To evaluate hepatic fibrosis progression or regression in CHC patients after sofosbuvir-based therapy.
2. To evaluate the durability of sustained viral response (SVR) in patients achieving SVR after sofosbuvir-based therapy.
3. To evaluate long-term effect of sofosbuvir-based therapy on the extra-hepatic manifestations of the cohort. The items include mixed cryoglobulinemia, chronic kidney diseases, insulin resistance, diabetic status, cardiovascular events and dyslipidemia.
4. To evaluate long-term effect of sofosbuvir-based therapy on quality of life on the cohort.

Study Design Prospective, longitudinal observational study

Study procedure A total of 200 patients receiving sofosbuvir based direct antiviral agents (DAAs) in the parent studies will be included for following up to 5 years. Their serological, image study and disease status description will be prospectively documented to present the long term effects of sofosbuvir-based therapy.

The presentation of illness will be specified as:

1. Main hepatic complications as liver fibrosis, hepatic malignancy, liver decompensation with ascites, hepatic encephalopathy and variceal bleeding, and liver-related mortality.
2. Life quality, extrahepatic symptoms as cryoglobulinemia, diabetes mellitus, insulin resistance, lipid profiles, renal insufficiency and other non-liver morbidities and malignancy.

ELIGIBILITY:
Main inclusion criteria:

For Sofosbuvir-based therapy observational group:

* Patients ≥ 20 of years who had ever participated in parent studies, GS-US-337-0131 (NCT02021656) or GS-US-334-0115 (NCT02021643)
* Patients who had received at least one dose of sofosbuvir-based therapy in the parent studies.

Who IFN-based therapy historical controls, matched with sex, age, level of liver fibrosis and virological response:

* Patients ≥ 20 of years who had received pegylated interferon plus ribavirin therapy with match of sex, age, level of liver fibrosis and virological response
* Patients who have ever participated study will be collected as historical control.

Main exclusion criteria:

* Patients not qualified by the main inclusion criteria were excluded.

For Sofosbuvir-based therapy observational group:

* Patients < 20 of years
* Patients who are unwilling to participate the current study
* Patients who had never participated in parent studies, GS-US-337-0131 (NCT02021656) nor GS-US-334-0115 (NCT02021643)
* Patients who had never received at least one dose of sofosbuvir-based therapy in the parent studies.

Who IFN-based therapy historical controls:

* Patients < 20 of years
* Patients who are unwilling to participate the current study
* Patients who had never received pegylated interferon plus ribavirin therapy
* Patients who did not participate study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had ever participated the parent studies, GS-US-334-0115 or GS-US-337-0131, will be invited to participate the current study in outpatient clinic. For the patients who have participated study will be invited to participate the current study as matched historical control n our outpatient clinic, Written informed consent will be obtained after full explanation to the patients who had ever participated in parent studies, GS-US-337-0131 (NCT02021656) or GS-US-334-0115 (NCT02021643) and had received at least one dose of sofosbuvir-based therapy in the parent studies.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with liver-related morbidity development during 5-year follow-up period after sofosbuvir-based treatment | 6 years
  Number of participants with liver-related morbidity during 5-year follow-up period after sofosbuvir-based treatment, including liver fibrosis progression and decompensation
Number of participants with liver-related mortality development during 5-year follow-up period after sofosbuvir-based treatment | 6 years
  Number of participants with liver-related mortality assessed by death due to HCC and/or liver decompensation
Number of participants with hepatocellular carcinoma (HCC) development during 5-year follow-up period after sofosbuvir-based treatment | 6 years
  Number of participants with HCC assessed by histocytology or positive dynamic image plus alpha fetoprotein (AFP) > 400 ng/ml

SECONDARY OUTCOMES:
Life quality | 6 years
  The change of short form(SF)-36 from baseline
Cryoglobulinemia | 6 years
  Change of proportion of participants with cryoglobulinemia from baseline cryoglobulinemia from baseline)
Diabetes mellitus (DM) | 6 years
  Number of participants without DM develop DM assessed by Ac sugar > 126 g/ml
Insulin resistance | 6 years
  Change of homeostatic model assessment (HOMA-IR), assessed by Glucose x insulin/22.5 from baseline
Lipid profiles | 6 years
  Change of the serum profile of lipids including triglyceride(TG), cholesterol(Chol), low-density lipoprotein-cholesterol (LDL-C), high-density lipoprotein-cholesterol (HDL-C) from baseline
Renal disease | 6 years
  the change of the estimated glomerular filtration rate (eGFR) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, Study Director — Kaoshiung Medical University Hospital; Chia-Yen Dai, Principal Investigator — Kaoshiung Medical University Hospital; Jee-Fu Huang, Principal Investigator — Kaoshiung Medical University Hospital; Chung-Feng Huang, Principal Investigator — Kaoshiung Medical University Hospital; Ming-Lun Yeh, Principal Investigator — Kaoshiung Medical University Hospital; Ching-I Huang, Principal Investigator — Kaoshiung Medical University Hospital; Ta-Wei Liu, Principal Investigator — Kaoshiung Medical University Hospital
Locations (26):
- South Korea (15):
  - Korea University Ansan Hospital, Ansan
  - Asan Medical Center, Asan
  - Soon Chun Hyang University Hospital Bucheon., Bucheon-si
  - Dong-A University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Gachon University Gil Hospital, Incheon
  - Pusan National University Hospital, Pusan
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hosptial, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Seoul
- Taiwan (11):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaoshiung Medical University Hospital, Kaohsiung City
  - Keelung Chang Gung Memorial Hospital, Keelung
  - China Medical University, Taichung
  - Chi Mei Liouying Hospital, Tainan
  - MacKay Memorial Hospital, Taipei
  - National Cheng Kung University Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CF, Heo J, Chien RN, Baek YH, Kao JH, Kim JH, Chang TT, Byun KS, Chen JJ, Jeong SH, Hu TH, Kim YS, Peng CY, Tak WY, Wang HY, Yoon SK, Sheen IS, Youn-Jae Lee, Hsu YC, Yim HJ, Tsai PC, Yeh ML, Ahn SH, Dai CY, Paik SW, Huang JF, Kim YJ, Chuang WL, Lim YS, Yu ML. Long-Term Hepatic and Extrahepatic Outcomes of Chronic Hepatitis C Patients After Sofosbuvir-Based Treatment (LONGHEAD Study). Infect Dis Ther. 2025 May;14(5):1089-1101. doi: 10.1007/s40121-025-01145-y. Epub 2025 Apr 10. PMID 40205145